CLINICAL TRIAL: NCT05099432
Title: The Cap-Assisted Resection Margin Assessment (CARMA) Technique After Polyp Resection: a Prospective Feasibility Study of a "Novel" Approach to Reduce Polyp Recurrence
Brief Title: The CARMA Technique Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Alexander Huelsen, Interventional Gastroenterologist, Principal Investigator, Princess Alexandra Hospital, Brisbane, Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 75076
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Colonic Polyp; Colonic Sessile Serrated Lesion
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARMA Technique (Experimental): All included participants undergo polyp resection using standard of care polypectomy techniques, followed by the CARMA technique
  Interventions: Procedure: CARMA technique

INTERVENTIONS:
Procedure: CARMA technique — Once standard polyp resection and assessment of the polypectomy site without magnification is completed, the CARMA technique will be applied. This will involve an assessment of the entire polypectomy margin using cap assisted magnification endoscopy with the ability to also use NBI (at the endoscopist's discretion) and documentation of any residual polyp noted.

SUMMARY:
Colonoscopic removal of polyps is an important and well-established tool in the prevention of colorectal cancers. However, high polyp recurrence rates after endoscopic resection, with resultant development of interval cancers, remains a problem; this most commonly stems from unrecognised incomplete polyp resection. Thus, a standardised endoscopic technique is needed that will allow endoscopists to consistently achieve a clear margin of resection. The investigators believe the Cap Assisted Resection Margin Assessment (CARMA) technique will address this problem. This novel technique focuses on a standardised assessment of the resection margin after endoscopic polypectomy utilising available standard high-definition video endoscopes with imaging features including narrow band imaging (NBI) and magnification endoscopy.

ELIGIBILITY:
Patients with colonic polyps will be considered following below criteria

Inclusion Criteria:

- any polypectomy (though only a maximum of two polyps from one individual participant)

Exclusion Criteria:

* polyps less than 10mm which were resected under endoscopic view with a definite > 1mm clear margin
* scar site recurrence polyps
* polyps with endoscopic evidence of invasion
* pedunculated polyps
* pseudopolyps
* participants who will not be available for follow up endoscopy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of achieving a clear resection margin using the CARMA technique | Established during index procedure

SECONDARY OUTCOMES:
Sensitivity and specificity of the CARMA technique for residual polyp detection | Established during index procedure
Frequency of residual polyp without CARMA assessment | Established during index procedure
Incomplete resection rate with use of CARMA technique | Established during index procedure
Incomplete resection rate with use of the CARMA technique in polyps > 10mm with hot snare | Established during index procedure
Incomplete resection rate with use of the CARMA technique in polyps > 10mm with cold snare | Established during index procedure
Residual polyp rate after CARMA technique with hot snare | Established during index procedure
Residual polyp rate after CARMA technique with cold snare | Established during index procedure
Time required for application of the CARMA technique with < 10mm | Established during index procedure
Time required for application of the CARMA technique with > 10mm | Established during index procedure
Polyp recurrence rate for < 10mm polyps | Established during surveillance procedure (following national guidelines - between 6 months to 5 years)
Polyp recurrence rate for > 10mm polyps | Established during surveillance procedure (following national guidelines - between 6 months to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Huelsen, MD, Principal Investigator — Princess Alexandra Hospital
Locations (1):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT05099432/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT05099432/ICF_001.pdf